CLINICAL TRIAL: NCT05201040
Title: A Prospective, Randomized, Evaluator/Subject-blinded, Double-Center, Controlled Clinical Study: Evaluate the Safety and Effectiveness of Mannitol-combined Hyaluronan Supplement in the Treatment of Knee Osteoarthritis.
Brief Title: Evaluate the Safety and Effectiveness of Mannitol-combined Hyaluronan Supplement in the Treatment of Knee OA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SciVision Biotech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RDCT-VSJK
Record Dates: First submitted 2022-01-05; First posted 2022-01-21 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-05

CONDITIONS: Knee Osteoarthritis; Hyaluronic Acid
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mannitol-combined Hyaluronic acid (Experimental): 2.0mL/syringe for one treatment
  Interventions: Device: JETKNEE Synovial Fluid Supplement
- Normal saline (Placebo Comparator): 2.0mL for one treatment
  Interventions: Device: Normal saline

INTERVENTIONS:
Device: JETKNEE Synovial Fluid Supplement — 2mL of JETKNEE Synovial Fluid Supplement
  Arms: Mannitol-combined Hyaluronic acid
Device: Normal saline — 2mL of normal saline
  Arms: Normal saline

SUMMARY:
To evaluate the effectiveness and safety of JETKNEE Synovial Fluid Supplement for alleviating pain of knee osteoarthritis (OA).

DETAILED DESCRIPTION:
The medical device is a bioabsorbable, extensible, crosslinked, 2% hyaluronic acid gel using micro-organism fermentation sourced hyaluronic acid as a major component and add mannitol is added which can inhibit the degradation of hyaluronate acid by free radicals to prolong the therapeutic effect. The medical device is injected into the articular cavity to protect joint tissue, increase joint lubricity, inhibit degradation of cartilage and promote the metabolism of cartilage by infiltrating degenerated cartilage. In addition, the medical device can penetrate the synovial tissue to inhibit inflammation and degradation. It also inhibits pain mediators in the synovium to achieve the pain inhibition. This study is to evaluate the effectiveness and safety of JETKNEE Synovial Fluid Supplement for alleviating pain of knee OA 6 months after single injection.

ELIGIBILITY:
Inclusion Criteria:

1. Age 45 to 85 years of male or female.
2. Meet the ACR diagnostic criteria, the target knee is confirmed with OA by radiographic images and Kellgren &Lawrence (K-L) score of 2 to 3；
3. Patients who still suffer from OA pain after receiving traditional non-drug therapy or general analgesic therapy within 6 months before the start of the study；
4. The VAS pain score of target knee must be at least 3 cm within 1 week before the screening and if the other side of knee has OA at the same time, the VAS pain score should be less than 3 cm；
5. Subject who has ability to understand the study purpose, comply with the study requirements, willing to stop all pain medications and physical therapy to the knees during the study and sign informed consent form (ICF).

Exclusion Criteria:

1. The hip or ankle joints are diagnosed with OA, pain, or deformity；
2. K-L score of 4 by radiographic image evaluation；
3. The target knee has symptoms such as infection, redness, and swelling at the screening period and before treatment ；
4. The target knee has received hyaluronic acid treatment within 6 months before included in the study；
5. The target side has received lower limb surgery or knee operation with accompanied complications and significant mobility impairment within 6 months before the start of the study；
6. The target knee has received treatments such as steroid injection, arthrocentesis or arthroscopic surgery within 3 months before screening；
7. Patient with autoimmune disease (such as autoimmune collagenopathy, rheumatoid arthritis), malignant tumors, coagulation disorder, heart diseases, mental diseases…etc. which may cause higher risk to patients during participation in the study；
8. Receiving orthopedic-related treatments which may affect the evaluation of the study；
9. With history of hypersensitivity or allergy to hyaluronic acid or any component of the device; With history of hypersensitivity or allergy to Gram-positive bacteria or Streptococcus proteins；
10. Pregnant, planning pregnancy or in breastfeeding females during the study period；
11. Subject who cannot cooperate with the follow- ups；
12. Other circumstances which judged to be unsuitable for participating in the study by the investigator.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
The pain score of Visual Analog Scale (VAS) of target knee at 6 months post-treatment. | 6 months post-treatment
  The pain score of Visual Analog Scale (VAS) of target knee at 6 months post-treatment.
  Based on the patient described pain intensity as 0 to 10 score, a higher score indicates greater pain intensity.

SECONDARY OUTCOMES:
The pain score of VAS of target knee at baseline, 2 weeks, 1 month, and 3 months post-treatment | baseline, 2 weeks, 1 month, and 3 months post-treatment
  The pain score of VAS of target knee at baseline, 2 weeks, 1 month, and 3 months post-treatment.
  Based on the patient described pain intensity as 0 to 10 score, a higher score indicates greater pain intensity.
The average score of Western Ontario and McMaster Universities (WOMAC) in pain section of the target knee at baseline, 2 weeks, 1 month, 3 months and 6 months post-treatment | baseline, 2 weeks, 1 month, 3 months and 6 months post-treatment
  The average score of Western Ontario and McMaster Universities (WOMAC) in pain section of the target knee at baseline, 2 weeks, 1 month, 3 months and 6 months post-treatment The WOMAC measures five items for pain (score range 0-20).Higher scores indicate worse pain, stiffness, and functional limitations.
The average score of WOMAC in stiffness section of target knee at baseline, 2 weeks, 1 month, 3 months and 6 months post-treatment | baseline, 2 weeks, 1 month, 3 months and 6 months post-treatment
  The average score of WOMAC in stiffness section of target knee at baseline, 2 weeks, 1 month, 3 months and 6 months post-treatment.
  The WOMAC measures two for stiffness (score range 0-8).Higher scores indicate worse pain, stiffness, and functional limitations.
The average score of WOMAC in function section of target knee at baseline and 2 weeks, 1 month, 3 months and 6 months post-treatment | baseline, 2 weeks, 1 month, 3 months and 6 months post-treatment
  The average score of WOMAC in function section of target knee at baseline and 2 weeks, 1 month, 3 months and 6 months post-treatment.
  The WOMAC measures 17 for functional limitation (score range 0-68).Higher scores indicate worse pain, stiffness, and functional limitations.
The average total score of WOMAC of the target knee at baseline, 2 weeks, 1 month, 3 months and 6 months post-treatment | baseline, 2 weeks, 1 month, 3 months and 6 months post-treatment
  The average total score of WOMAC of the target knee at baseline, 2 weeks, 1 month, 3 months and 6 months post-treatment.
  The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68).Higher scores indicate worse pain, stiffness, and functional limitations.
The average total score of Lequesne's Index (LI) of target knee at baseline and 2 weeks, 1 month, 3 months and 6 months post-treatment | baseline and 2 weeks, 1 month, 3 months and 6 months post-treatment
  The average total score of Lequesne's Index (LI) of target knee at baseline and 2 weeks, 1 month, 3 months and 6 months post-treatment
The thickness of femoral Intercondylar cartilage of the target knee by ultrasound at baseline, 1 month, 3 months and 6 months post-treatment | baseline and1 month, 3 months and 6 months post-treatment
  The thickness of femoral Intercondylar cartilage of the target knee by ultrasound at baseline, 1 month, 3 months and 6 months post-treatment
The quadriceps thickness of the target knee by ultrasound at baseline and 1 month, 3 months and 6 months post-treatment | baseline and 1 month, 3 months and 6 months post-treatment
  The quadriceps thickness of the target knee by ultrasound at baseline and 1 month, 3 months and 6 months post-treatment
The grade of cartilage of target knee by ultrasound at baseline, 1 month, 3 months and 6 months post-treatment | baseline, 1 month, 3 months and 6 months post-treatment
  The grade of cartilage of target knee by ultrasound at baseline, 1 month, 3 months and 6 months post-treatment
Holding time of Single-leg Stance Test (SLS) on target knee at baseline and 2 weeks, 1 month, 3 months and 6 months post-treatment | baseline and 2 weeks, 1 month, 3 months and 6 months post-treatment
  Holding time of Single-leg Stance Test (SLS) on target knee at baseline and 2 weeks, 1 month, 3 months and 6 months post-treatment
Subject self-evaluating satisfaction at 2 weeks, 1 month, 3 months and 6 months post-treatment | 2 weeks, 1 month, 3 months and 6 months post-treatment
  Subject self-evaluating satisfaction at 2 weeks, 1 month, 3 months and 6 months post-treatment

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Kaohsiung Municipal Siaogang Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City

IPD SHARING:
Plan to Share IPD: No